CLINICAL TRIAL: NCT07024069
Title: Tongue Shear-wave Elastography and Attenuation Ultrasound Markers in Healthy Subjects: a Protocol Study
Brief Title: Protocol for Tongue Elastography and Ultrasound Markers
Status: Completed | Type: Observational
Sponsor: Haute Ecole Bruxelles-Brabant (Other)
Responsible Party: Principal Investigator, Frédéric Paillaugue, Principal Investigator, MSc PT Drs, Haute Ecole Bruxelles-Brabant
Other Study IDs: B200-2024-057
Record Dates: First submitted 2025-05-28; First posted 2025-06-17 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Healthy Individuals (Controls)
Keywords: tongue ultrasound; submental ultrasound; tongue stiffness; echo intensity
MeSH Terms: interventions — Weights and Measures; Body Height

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adult subjects: Healthy subjects (aged 18-45), male and female. All subjects will give their informed consent. Consequently, exclusion criteria will include any orthopaedic, traumatological or rheumatic pathology of the cervico-cephalic extremities, as well as any metabolic (diabetes, metabolic syndrome, etc.) or cardiovascular pathology. In particular, subjects must not suffer from sleep disorders or OSA, as identified by the Berlin Sleep Questionnaire and Stop-BANG questionnaire. Subjects will be asked not to consume alcohol or drugs 48 hours before the experiment.
  Interventions: Other: Tongue ultrasound via submental approach

INTERVENTIONS:
Other: Tongue ultrasound via submental approach — Descriptive and anthropometric data will be recorded for each participant, including age, sex, weight (kg), height (m), neck circumferences (cm). Body mass index (expressed in kg/m2) will be calculated.
  Submental ultrasound (US) images of the tongue will be performed on a patient lying supine, using a 5-15 MHz convex transducer. The parameters will be identical for all subjects and set at a depth of 9 cm, a focus of 4 cm and a gain of 45%. Each measurement will be taken thrice by a trained operator; the mean and standard deviation being used for analysis.
  Other Names: Weight, height, neck circumference

SUMMARY:
The purpose of this observational is to methodologically assess the standardisation and reliability of a protocol of ultrasound lingual markers, including tongue shear-wave elastography, attenuation indexes, and echo intensity in adult healthy subjects.

The main goals are to create a standardized protocol and its intra- et inter-rater reliability, in order to gather some data in a non-pathological population. This protocol will be used in further studies in the context of tongue fat accumulation, such as in obstructive sleep apnea syndrome.

Participants will be lying in supine position and after basic descriptive data collection (height, weight, neck circumference), submental ultrasound will be performed on them. This procedure is non-invasive, painless, safe (ultrasound does not involve ionising radiation) for the healthy participants.

DETAILED DESCRIPTION:
Scientific literature is reporting increasing evidence that fat accumulation in the tongue and oropharyngeal region is linked to cardiovascular disorders in people with obesity. In this context, fat accumulation on the tongue is a contributing factor to Obstructive Sleep Apnea syndrome (OSA). The presence of OSA is a significant risk factor for the development of cardiovascular disease and is directly correlated with overall adiposity, while the percentage of neck fat relative to the abdomen is correlated with the severity of OSA in obese individuals, highlighting the relevance of studying body fat distribution. The links between increased tongue size, neck and oropharyngeal adiposity, BMI, and sleep-disordered breathing have been supported by magnetic resonance imaging (MRI) and cone beam computed tomography studies and are now well documented. It is interesting to note that OSA also affects people who are not obese, highlighting the relevance of studying its risk factors. Excessive lipid accumulation in peripheral tissues therefore appears to be a key feature of many metabolic diseases. Thus, early detection of excessive lipid accumulation in tissues and therapeutic monitoring are key to prevention and individualised, patient-centred care. Ultrasound has recently been used to establish a link between oropharyngeal fat and OSA: studies showed that changes in the dynamic properties of the tongue muscles measured by elastography, or the size and volume of the tongue, could be a biomarker for screening for OSA in adults. Shear wave elastography (SWE) is already used for fat accumulation in various organs, for example in liver or kidney diseases, and some authors have begun to work on the musculoskeletal system. This technique uses acoustic force to generate shear waves (which can propagate perpendicular to the ultrasound beam, causing transient tissue deformation that can be measured by the machine's module), providing a measure of the elastic properties of the tissue, which is reported as 'rigidity' or 'stiffness'. When muscles are infiltrated by lipid deposits, the histological content changes, leading to a modification of tissue properties. This ultrasound approach is a simple, non-irradiating and harmless technique that could be applied in the future therapeutic follow-up of patients with OSA.

Moreover, it is important to underscore that the lingual ultrasound markers analysed in this study are not solely indicative of fat content within the tongue. They are also likely to depict biomechanical characteristics of tongue tissues. Indeed, these markers can be influenced by various compositional and structural changes, including modifications in fat content, connective or fibrous tissue density, presence of edema or swelling... As such, variations in ultrasound-derived parameters may determine a range of tissue properties beyond adiposity, providing a more comprehensive insight into the biomechanical state of the tongue that is particularly involved in obstructive sleep apnea. This lingual ultrasound protocol could then be use in further studies by applying it in patients suffering from OSA.

Study objectives: The main objective of this study is to investigate ultrasound markers of fat accumulation in the tongue in healthy individuals, to assess the reliability and repeatability of the measurement, and to determine the distribution of tongue fat values in different regions of the tongue. The secondary objective will be to study the correlations of these values with the subjects' basic anthropometric data. The aim of obtaining values in healthy subjects will be to compare them with a future study on a population suffering from OSA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-45 years
* Able to understand and provide informed consent

Exclusion Criteria:

* Any orthopaedic, traumatic, or rheumatic conditions affecting the head or neck
* Presence of metabolic disorders (e.g., diabetes, metabolic syndrome)
* Presence of cardiovascular conditions
* Diagnosed sleep disorders or known sleep apnea syndrome, as evaluated by the Stop-Bang and Berlin questionnaires
* Consumption of alcohol or drugs within 48 hours prior to the experiment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects (aged 18-45), male and female, recruited from physiotherapy students at ISEK-HE2B and health students at VUB (Brussels Health Campus site in 1090 Jette) and their relatives.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Tongue stiffness (ultrasound) | Day 1
  Tongue stiffness (in kPa), measured with shear-wave elastography (ultrasound submental approach)
Tongue Echo Intensity (ultrasound) | Day 1
  Tongue Echo Intensity, expressed as the mean value of pixels in a 0-255 gray scale (ultrasound submental approach)
Tongue Tissue Attenuation Imaging (ultrasound) | Day 1
  Tongue Tissue Attenuation Imaging, measured with ultrasound submental approach, reflecting the quantitative measurement of US attenuation in tissue in dB/cm/MHz
Tongue thickness (ultrasound) | Day 1
  Tongue thickness (in cm, measured via ultrasound submental approach), reflects its size, representing the vertical distance between its most superior surface point to its most inferior

SECONDARY OUTCOMES:
Age | Day 1
  Age (in years) will be collected via a questionnaire
Weight | Day 1
  Weight (in kg) will be measured with a weighing scale
Height | Day 1
  Height (in m) will be collected with a stadiometer
Neck circumference | Day 1
  Neck circumference (in cm) will be measured with a lufkin tape according to the International Society for the Advancement of Kinanthropometry (ISAK) guidelines.
Body Mass Index (BMI) | Day 1
  Weight and height will be combined to report BMI in kg/m^2

OTHER OUTCOMES:
Berlin Sleep Questionnaire | Day 1
  The Berlin Sleep questionnaire consists of 3 categories relating the risk of suffering from sleep apnea.
Stop-Bang Questionnaire | Day 1
  The STOP-BANG questionnaire screens for obstructive sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Steven Provyn, PhD, Study Director — HE2B & VUB
Locations (1):
- Isek He2B, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided